CLINICAL TRIAL: NCT05571735
Title: Immunogenicity of COVID-19 Vaccines Against Coronavirus Disease (COVID-19) Among Tuberculosis (TB) Patients in Thailand-Myanmar Border.
Brief Title: Immunogenicity of COVID-19 Vaccines in Tuberculosis Patients
Acronym: CVTB
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: VIR21002
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Covid-19 Pandemics; Tuberculosis
MeSH Terms: conditions — COVID-19; Tuberculosis | interventions — BNT162 Vaccine; ChAdOx1 nCoV-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Leftover blood specimens will be stored for possible confirmatory or additional testing. In the event that the stored specimen is used for purposes that may or may not be related to this study. SMRU will be responsible for obtaining the necessary ethical approvals. Samples stored for future use will be anonymized using a standard operating procedure (SOP) and coded so that no identification of the subject is possible. Stored samples will be destroyed after a maximum of 10 years after study close. Sample disposal will be done as per related SOPs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TB cohort: TB cohort - Bacteriologically confirmed TB patients (18 years and above)
  One of the following three COVID-19 vaccines will be provided based on availability of supply from the Ministry of public health, Thailand as an intervention for the study.
  Interventions: Biological: Pfizer-BioNTech COVID-19 vaccine; Biological: AstraZeneca vaccine; Biological: Janssen Ad26.COV2.S COVID-19 vaccine
- Healthy comparator: Comparator- Clinically healthy individuals (54 in healthy comparator)
  One of the following three COVID-19 vaccines will be provided based on availability of supply from the Ministry of public health, Thailand as an intervention for the study.
  Interventions: Biological: Pfizer-BioNTech COVID-19 vaccine; Biological: AstraZeneca vaccine; Biological: Janssen Ad26.COV2.S COVID-19 vaccine

INTERVENTIONS:
Biological: Pfizer-BioNTech COVID-19 vaccine — Pfizer-BioNTech COVID-19 vaccine, Messenger RNA (mRNA) based vaccine encoding the viral spike glycoprotein (S) Formulation: Frozen concentrate before dilution with 0.9% sodium chloride solution for injection Route of Administration: Intramuscular (IM) Dosing regimen: Two doses (0.3 mL per dose) (at least 3 weeks apart)
Biological: AstraZeneca vaccine — AstraZeneca vaccine, a replication-deficient simian adenoviral vector expressing the spike (S) protein of SARS-CoV-2 Formulation: Aqueous solution for injection Route of Administration: Intramuscular (IM) Dosing regimen: Two doses (0.5 mL per dose) (at least 12 weeks apart)
Biological: Janssen Ad26.COV2.S COVID-19 vaccine — Janssen Ad26.COV2.S COVID-19 vaccine, recombinant, replication-incompetent adenovirus serotype 26 (Ad26) vector encoding a full-length and stabilized SARS-CoV-2 spike protein.
  Formulation: Suspension for injection Route of Administration: Intramuscular (IM) Dosing regimen single dose (0.5 mL)

SUMMARY:
This study is a non-randomized observation and comparison of immune response between bacteriologically confirmed TB patients under treatment cohort who received COVID-19 vaccine (n=54) vs healthy individuals (n=54).

Each participant will receive single or double doses of one of COVID-19 vaccines (Pfizer-BioNTech COVID-19 vaccine, AstraZeneca vaccine or Janssen Ad26.COV2.S COVID-19 vaccine) in the deltoid muscle of the non-dominant arm. Study Duration approximately 1 year. The main focus of this study is to compare the humoral and cellular immunological responses of the COVID-19 vaccines between bacteriologically confirmed TB patients under treatment vs healthy individuals.

This study is funded by the Wellcome Trust. The grant reference number is 220211/A/20/Z.

DETAILED DESCRIPTION:
In late 2020, COVID-19 pandemic was occurred globally. Like Tuberculosis (TB), severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection is primarily affected in respiratory tract with increased risk of severe clinical complications especially in particular risk population like diabetic patients and old ages. Like other viral infections, there is evidence that both acquired humoral and cellular immunological responses against the SARS-CoV-2 infection are key in providing protective immunity. Although the magnitude and durability of both binding and neutralizing antibodies after seroconversion of COVID-19 patients are highly variable at the individual patient level, higher level of neutralizing antibodies appears to be correlated with protection against reinfection.

As natural immunity alone after COVID-19 infection appears to be insufficient for protection against COVID-19, since the beginning of COVID-19 pandemic, several COVID-19 vaccines developed based on different technical platforms have been introduced globally. Up to August 2021, twenty COVID-19 vaccines has been included in WHO's Emergency Use Listing (EUL).

As protection against COVID-19 infection among TB patients is critical to prevent severe clinical outcomes, COVID-19 immunization program is carrying out among TB patients in the SMRU TB centers with supply of COVID-19 vaccines from Ministry of public health, Thailand. In Thailand, Pfizer-BioNTech COVID-19 vaccine, AstraZeneca vaccine and Janssen Ad26.COV2.S COVID-19 vaccine are widely available in COVID-19 vaccination campaigns.

Pfizer-BioNTech COVID-19 vaccine is an mRNA vaccine and its two-dose regimen with inter-dose interval of 21 days apart can provide effective protection against SARS-CoV-2- infection. Mild local and systemic reactions can occur after vaccination but serious adverse effects can be complicated rarely. It can also be provided for children over 6 months of age and reactogenicity is also less frequent.

AstraZeneca vaccine is a replication-deficient chimpanzee adenovirus-vectored vaccine expressing full-length SARS CoV-2 spike glycoprotein gene. Efficacy, immunogenicity and safety profiles of the vaccine are acceptable and reasonably well tolerated in healthy young and old adults, symptomatic COVID-19 patients and people with HIV infection.

Janssen Ad26.COV2.S COVID-19 vaccine is a recombinant, replication-incompetent adenovirus serotype 26 (Ad26) vector encoding a full-length and stabilized SARS-CoV-2 spike protein. The vaccine needs single dose of administration intramuscularly into the deltoid muscle. Multicenter, placebo-controlled, phase 1-2a trial has shown that single dose of the vaccine has an efficacy of 66.9% against symptomatic COVID-19 infection, 76.7% against severe COVID-19 disease after 14 days, and 85.4% after 28 days. The vaccine appears to be safe like other COVID-19 vaccines because no severe allergic or anaphylactic reaction has been recorded in clinical trials except from occurrence of a very rare syndrome of blood clotting combined with low platelet counts in some countries. However, there has been no sufficient data on pregnancy and people with co-morbidity especially HIV/TB patients.

As there is limited knowledge about immunogenicity of COVID-19 vaccines among TB patients, examination of immunological responses from the COVID-19 vaccines offering in community COVID-19 vaccination campaigns among TB patients as well as healthy population is warranted. Protectability and immune response to the COVID-19 vaccines in TB patients under treatment should be studied to get better understanding about immunological responses among population with co-morbidity. Along with antibodies response, reactogenicity, clinical and laboratory safety profiles of the COVID-19 vaccines in this specific group will also be assessed and compared with the healthy control.

This study is a non-randomized observational study aimed to compare humoral and cellular immunological responses of the COVID-19 vaccines between bacteriologically confirmed TB patients under treatment cohort (n=54) vs healthy individuals (n=54) after receiving a COVID-19 vaccine. Each participant will receive single or double doses of one of aforementioned COVID-19 vaccines in the deltoid muscle of the non-dominant arm.

Follow-up appointments will be scheduled on 2nd dose visit and 28 days after 2nd dose in double dose scheduled COVID-19 vaccines and 28 days and 56 days after vaccination in single dose scheduled COVID-19 vaccine. For assessment of reactogenicity, participants will be informed to attend follow-up appointments every day for 7 days following each dose of vaccination.

Frequency, incidence and nature of solicited local and systemic adverse events (AEs) and unsolicited AEs will be recorded at their follow up visits. For immunological responses, humoral and cellular antibody level to SARS-CoV-2 virus will be assessed over time (before 1st dose, before 2nd dose , 28 days after 2nd dose in double dose scheduled COVID-19 vaccine or before single dose vaccination, 28 days and 56 days after vaccination in single dose scheduled COVID-19 vaccine) and compared between TB patients and healthy individuals. Baseline laboratory investigations such as liver function tests, renal function tests, serum electrolytes, iron, complete blood count and C reactive protein will be tested on Day 0 and rechecked on the same days as immunological tests to review changes after vaccination.

Infection serological tests such as Human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), and Hepatitis C antibody (HCV Ab) tests will be performed at screening visit with consent of potential participants. Moreover, nasopharyngeal swab for COVID-19 PCR test will be tested before being enrolled. These tests can be repeated if there are symptoms suggestive of these infections.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above, newly diagnosed bacteriologically confirmed TB patients including both drug sensitive and resistant TB, who are taking anti TB or MDR-TB treatment in initial period during study period or clinically healthy individuals for comparator arm.
* Willing to be followed for four weeks following second dose of Pfizer-BioNTech COVID-19 vaccine and AstraZeneca vaccine or eight weeks following single dose of Janssen Ad26.COV2.S COVID-19 vaccine
* Willing to be involved in the pre-enrolment screening.
* For women with child bearing potential only (aged 18-49 years), willing to continue to use effective contraception methods through the study.
* For women with child bearing potential only (aged 18-49 years), negative pregnancy test on the day of screening and on the day of vaccination to be eligible to receive the vaccination.
* Able and willing to comply with all study requirements.
* Ability to understand the study instructions and provide written informed consent

Exclusion Criteria:

* History of laboratory confirmed COVID-19 for any duration before or positive COVID-19 PCR or antigenic test at screening.
* History of HIV infection
* Participation in other COVID-19 related studies for the duration of the study.
* Participation in other vaccine trials within 90 days before and 30 days after the study vaccination.
* Administration of any immunoglobulins or any type of COVID-19 vaccine within 90 days before administration of the vaccine.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any previous history of a serious side effect with any kind of vaccine.
* Any history of angioedema.
* Any history of anaphylaxis.
* Women with pregnancy, lactation or planning to get pregnant during the duration of the study.
* Current diagnosis of or treatment for cancer.
* History of severe psychiatric disorders likely to affect participation in the study.
* Bleeding disorder (e.g. coagulation factor deficiency, coagulopathy or platelet disorder), history of thrombosis or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Suspected or known current alcohol or drug dependency (except well controlled condition).
* Presence of any condition which in the judgement of the investigator would place the patient at undue risk or interfere with the results of the study.
* Severe and/or uncontrolled cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well controlled comorbidities are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TB cohort - Bacteriologically confirmed TB patients (54 in cohort of patients)
  Comparator- Clinically healthy individuals (54 in healthy comparator)
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of humoral and cellular responses to SARS-CoV-2 between bacteriologically confirmed TB patients under treatment vs healthy individuals at the end of the study | Day 49 in Pfizer-BioNTech COVID-19 vaccine, Day 112 in AstraZeneca vaccine or Day 56 in Janssen Ad26.COV2.S COVID-19 vaccine
Comparison of humoral and cellular responses to SARS-CoV-2 between bacteriologically confirmed TB patients under treatment vs healthy individuals. | Day 21 in Pfizer-BioNTech COVID-19 vaccine, Day 84 in AstraZeneca vaccine or Day 28 in Janssen Ad26.COV2.S COVID-19 vaccine

SECONDARY OUTCOMES:
Occurrence and comparison of solicited local reactogenicity signs and symptoms for 7 days following each dose of vaccination | 7 Days
Occurrence and comparison of solicited systemic reactogenicity signs and symptoms for 7 days following each dose of vaccination | 7 Days
Occurrence and comparison of unsolicited adverse events (AEs) following each dose of vaccination | Day 0, Day 7, Day 21, Day 28, Day 49, Day 56, Day 84, Day 112 in each vaccination
  Day 0, 7 days following first dose of vaccination, Day 21, 7 days following second dose of vaccination, Day 49 in Pfizer-BioNTech COVID-19 Vaccine, Day 0, 7 days following first dose of vaccination, Day 84, 7 days following second dose of vaccination, Day 112 in AstraZeneca vaccine or Day 0, 7 days following single dose of vaccination, Day 28 and Day 56 in Janssen Ad26.COV2.S COVID-19 vaccine
Comparison of changes from baseline for safety laboratory measures between bacteriologically confirmed TB patients under treatment vs healthy individuals. | Day 0, Day 21, Day 28, Day 84
  Comparison of changes from baseline for safety laboratory measures between bacteriologically confirmed TB patients under treatment vs healthy individuals at the day of second dose vaccination in double dose scheduled COVID-19 vaccine or 28 days following single dose of vaccine and the final day of study.

CONTACTS AND LOCATIONS:
Overall Officials: François Nosten, Professor, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Ramat, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All personal details of participants will be de-identified. These data including laboratory investigation results will be stored and may be shared to other researchers to apply in their research in accordance with the MORU data sharing policy.
Supporting Information: Study Protocol